CLINICAL TRIAL: NCT02457806
Title: Phase 1, Randomized, Double-Blind, Placebo-Controlled, 4-Period, Complete Cross-Over Comparison of the Anesthetic Efficacy of Bilateral and Unilateral Application of Kovacaine Mist in Healthy Volunteers
Brief Title: Comparison of Anesthetic Efficacy of Bilateral and Unillateral Application of Kovacaine Mist in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St. Renatus, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: SR 2-04
Record Dates: First submitted 2015-05-21; First posted 2015-05-29 (Estimated); Last update posted 2016-11-10 (Estimated); Status verified 2016-11

CONDITIONS: Anesthesia
Keywords: Dental Anesthesia
MeSH Terms: interventions — Tetracaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Kovacaine Mist (Experimental): 3 sprays of Kovacaine Mist (Tetracaine HCl 3% and Oxymetazoline HCl 0.05%) in each nostril (bilateral dosing) administered 4 minutes apart
  Interventions: Drug: Tetracaine HCl 3% and Oxymetazoline HCl 0.05%
- Kovacaine Mist and Placebo (Active Comparator): 3 sprays of Kovacaine Mist (Tetracaine HCl 3% and Oxymetazoline HCl 0.05%) in the right nostril and three sprays of placebo in the left nostril (right-sided unilateral dosing) administered 4 minutes apart
  Interventions: Drug: Tetracaine HCl 3% and Oxymetazoline HCl 0.05%; Drug: Placebo spray
- Placebo and Kovacaine Mist (Active Comparator): 3 sprays of Kovacaine Mist (Tetracaine HCl 3% and Oxymetazoline HCl 0.05%) in the left nostril and 3 sprays of placebo in the right nostril (left-sided dosing) administered 4 minutes apart
  Interventions: Drug: Tetracaine HCl 3% and Oxymetazoline HCl 0.05%; Drug: Placebo spray
- Placebo spray (Placebo Comparator): 3 sprays of placebo in each nostril administered 4 minutes apart
  Interventions: Drug: Placebo spray

INTERVENTIONS:
Drug: Tetracaine HCl 3% and Oxymetazoline HCl 0.05% — Active Spray with deliverable volume of 0.1 mL
  Other Names: Kovacaine Mist
  Arms: Kovacaine Mist; Kovacaine Mist and Placebo; Placebo and Kovacaine Mist
Drug: Placebo spray — Aqueous solution to deliver 0.1 mL per unit
  Other Names: Placebo
  Arms: Kovacaine Mist and Placebo; Placebo and Kovacaine Mist; Placebo spray

SUMMARY:
To compare the efficacy of Kovacaine Mist administered bilaterally to that of Kovacaine Mist administered unilaterally with respect to global profound pulpal anesthesia in target teeth numbers 4-13.

DETAILED DESCRIPTION:
Qualified and consenting healthy subjects will be randomly assigned in a double-blind manner to sequences of four randomly ordered study periods with inter-treatment "washout" periods of 3 to 14 days. The four study regimens, which will be applied in random order will be:

* Regimen1. Three sprays of Kovacaine Mist in each nostril (bilateral dosing);
* Regimen 2. Three sprays of Kovacaine Mist in the right nostril and three sprays of placebo in the left nostril (right-sided unilateral dosing);
* Regimen 3. Three sprays of Kovacaine Mist in the left nostril and three sprays of placebo in the right nostril (left-sided unilateral dosing);
* Regimen 4. Three sprays of placebo in each nostril (placebo dosing).

During each testing period, eight representative maxillary teeth (#s 3, 4, 6, 8, 9, 11, 13 and 14) will be assessed for anesthesia using standard EPT testing. EPT testing will be conducted on the eight representative teeth at the following time points (minutes relative to the first spray of study drug): T-5, T3, T7, T11, T16, T21, T26T31, T41, T51, T61, T76, T91, T121, T151, and T181. If EPT testing of a target tooth is not possible (e.g., missing or does not meet inclusion criterion #2) tooth substitution is permissible. For molar teeth, #2 may replace #3 and #15 may replace #14. For premolar teeth, #5 may replace #4 and #12 may replace #13. The same replacements will be made for all testing sessions, and the actual teeth tested will be documented in the CRF.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 years of age or older.
* Eight representative maxillary teeth [(3 (or 2), 4 (or 5), 6, 8, 9, 11, 13 (or 12), and 14 (or15)] free of observable decay (or other pathology), crowns or veneers, all of which have EPT values of 10-50 at screening.
* Normal lip, nose, eyelid, palate, and cheek sensation.
* Patency of both left and right nasal airways.
* Ability to understand and willingness to sign the study informed consent form, communicate with study investigators, and understand and comply with the requirements of the study protocol.

Exclusion Criteria:

* Poorly controlled hypertension (blood pressure greater than 150/90 mmHg) or history of coronary heart disease.
* Diabetes mellitus.
* Any active thyroid disease other than S/P thyroidectomy on thyroid hormone replacement with TSH values in the normal range.
* History or presence of narrow-angle glaucoma.
* Prostatic enlargement.
* History of sinus/nasal surgery that, in the opinion of the investigator, could confound study results.
* History of frequent nose bleeds.
* Receipt of dental care requiring a local anesthetic within the last 24 hours.
* History of allergy to or intolerance of tetracaine, benzyl alcohol, benzocaine, other ester local anesthetics, succinylcholine, or para-aminobenzoic acid (as found in PABA-containing sunscreens).
* History of allergy or hypersensitivity to articaine, oxymetazoline, epinephrine, or sulfite antioxidants.
* History of drug abuse.
* Use of a monoamine oxidase inhibitor within the 3 weeks immediately prior to anticipated study participation.
* Nursing, pregnant, suspected of being pregnant, or trying to become pregnant. (Females will be required to undergo pregnancy testing to rule out pregnancy)
* Use of any investigational drug and/or participation in a clinical research trial within 30 days of the first study dosing day.
* Requirement for uninterrupted use of any medication with actions that might, in the opinion of the involved investigator, confound interpretation of study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2011-08; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Achievement of GPPA by teeth reaching an EPT of 80 | 20 minutes of final spray
  Achievement of Global Profound Pulpal Anesthesia (GPPA) as having all three target maxillary teeth [nos. 4(or 5), 6, and 8 for the right side or nos. 9, 11, and 13 (or 12) for the left-side] reach an EPT of 80 within 20 minutes of the final spray of study drug

SECONDARY OUTCOMES:
Incidence of GPPA for bilateral versus placebo administration | 20 minutes of final spray
Incidence of PPA for individual teeth | 181 minutes
  For all individually EPT-tested teeth the incidence of Profound Pulpal Anesthesia (PPA) defined as reaching an EPT of 80 within 20 minutes, with unilateral and bilateral drug administration
Time to onset and duration of PPA | 181 minutes
  For all individually EPT-tested teeth achieving PPA, time to onset and duration of PPA for unilateral and bilateral drug administration
Mean highest EPT value reached for first molars (#3 and 14) | 181 minutes
Incidence of induction of PPA following the first, second and third doses of active drug administered unilaterally and bilaterally | 181 minutes
Correlation between positive responses on Subjective Numbness Assessment (DNA) and incidence of global EPT scores of 80 | 181 minutes
Systolic Blood Pressure | 181 minutes
Diastolic Blood Pressure | 181 minutes
Heart Rate | 181 minutes
Adverse experiences spontaneously reported | 24 hours
  Adverse experiences spontaneously reported by subjects, or observed by study personnel including those encountered on nasal and airway examination (NAE), incidence rates for systolic and diastolic blood pressure and heart rate exceeding +/- 25% of pre-study values

CONTACTS AND LOCATIONS:
Overall Officials: Patrick R Brain, DDS, Principal Investigator — Jean Brown Research
Locations (1):
- Jean Brown Research, Salt Lake City, Utah, United States